CLINICAL TRIAL: NCT06588348
Title: Corticosteroid Effect on Achalasia Variant Esophagogastric Junction Outflow Obstruction
Brief Title: Corticosteroid Effect on Achalasia Variant EGJOO
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Principal Investigator, Chanakyaram Reddy, Principle Investigator, Baylor Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 022-001 Steroid Study
Record Dates: First submitted 2024-08-23; First posted 2024-09-19 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Esophagogastric Junction Outflow Obstruction
Keywords: EGJOO; Corticosteroid
MeSH Terms: interventions — Prednisone; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Steroid Treatment (Experimental): All participants are in the treatment arm. Patients with Esophagogastric Junction Outflow Obstruction (EGJOO) will undergo steroid treatment for 14 days. On the last day of the 14 day treatment, patient will undergo esophageal manometry testing to assess for treatment response. They will also be asked to complete follow-up Eckardt and BEDQ surveys.
  Interventions: Drug: Steroid treatment; Procedure: Esophageal Manometry; Other: Survey

INTERVENTIONS:
Drug: Steroid treatment — All enrolled subjects will be prescribed a 14-day course of corticosteroid therapy in the form of Prednisone 20 mg to be taken once daily by mouth.
  Other Names: Prednisone
Procedure: Esophageal Manometry — On the final day of Prednisone use, all subjects will undergo esophageal manometry testing to assess for treatment response.
Other: Survey — All enrolled subjects will be asked to complete follow-up Eckardt and BEDQ surveys.
  Other Names: Eckardt and Brief Esophageal Dysphagia Questionnaire (BEDQ)

SUMMARY:
EGJOO is a disorder in which the muscles of the esophagus (swallowing tube) do not function in a coordinated fashion so that swallowed material does not pass easily into the stomach. EGJOO often causes symptoms of swallowing difficulties and chest pain. The cause of EGJOO and its optimal treatment are not clear. The investigators research team suspects that EGJOO might be caused by an allergy that involves the esophagus, and that treatment with medications called corticosteroids might improve function of the esophageal muscles. The purpose of this study is to learn how corticosteroid therapy affects the muscles of the esophagus in patients suffering with EGJOO.

DETAILED DESCRIPTION:
Esophagogastric junction outflow obstruction (EGJOO) is an esophageal motility disorder with a heterogeneous etiology. The optimal treatment for EGJOO is not known, and proper management of the condition remains disputed. Similar to patients with achalasia, patients with EGJOO exhibit poor relaxation of the lower esophageal sphincter (LES) with swallowing. Unlike patients with achalasia, however, those with EGJOO have some intact peristalsis in the esophageal body. Achalasia treatments (pneumatic dilation, Heller myotomy, per-oral endoscopic myotomy [POEM]) attempt to destroy LES muscle contraction function with myotomy inflicted by balloon distention (pneumatic dilation), diathermic needle-knife (POEM), or scalpel (Heller myotomy). With POEM and Heller myotomy, the incision extends into muscle of the esophageal body. These same interventions have been used to treat EGJOO, but an effective, non-invasive therapy that does not involve muscle disruption would be preferable, especially since EGJOO patients have evidence of esophageal body peristalsis that might be destroyed by achalasia myotomy techniques. The investigators Center for Esophageal Diseases has recently described a possible allergic etiology for achalasia and EGJOO in a study in which the investigators found profound mast cell degranulation in the LES muscle in all of 13 patients with these disorders who were treated with Heller myotomy. The investigators have also published reports outlining the investigators rationale for considering an allergic etiology for achalasia and EGJOO. Now, an extension of this work is to assess whether corticosteroid therapy, which can improve allergic conditions, can correct the esophageal dysfunction in EGJOO to the point that invasive and irreversible myotomy treatments might not be required. The proposed study will enroll subjects with clinically significant EGJOO on the achalasia-variant spectrum, and treat them with a 14-day course of oral, systemic corticosteroid therapy. The investigators aim to describe the symptomatic and manometric response to corticosteroid therapy, and hypothesize that the investigators findings might establish that a subset of patients with EGJOO have a reversible form of esophageal muscle dysfunction. Although long-term treatment with corticosteroids has unacceptable toxicity, identification of a reversible form of EGJOO with a short course of steroid therapy would suggest a therapeutic role for other, less toxic, allergy-directed therapies.

ELIGIBILITY:
Inclusion Criteria: Adult patients age 18 years or older with the following clinical and diagnostic criteria will be eligible for study inclusion:

* EGJOO manometric diagnosis based on CC v4.0 criteria
* Primary symptom of dysphagia and/or non-cardiac chest pain
* Additional objective evidence of obstruction on Timed Barium Esophagram and/or EndoFLIP
* The treating physician has determined that invasive therapy (botulinum toxin injection, pneumatic dilation, POEM, or Heller myotomy) is indicated.

Exclusion Criteria:

* History of prior foregut surgery
* History of esophageal botulinum toxin injection within 6 months of study enrollment
* Presence of hiatal hernia > 2 centimeters
* Presence of esophageal mass
* Obstructing esophageal stricture or ring on endoscopy
* Reflux esophagitis (LA Grades B-D)
* Subjects on current immunosuppression or immune modulating therapy
* Chronic opioid use
* Previously diagnosed extrinsic compression of the gastroesophageal junction
* Concomitant Eosinophilic Esophagitis with uncontrolled mucosal disease who have not tried at least one standard therapy
* Contraindication to the use of oral corticosteroids
* History and/or current diagnosis of Diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-07-26 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Response in esophageal motility to study intervention | Assessed upon being on study intervention medication for 14 days
  Median integrated relaxation pressure (IRP) of the lower esophageal sphincter (LES) obtained through esophageal manometry procedure

CONTACTS AND LOCATIONS:
Overall Officials: Chanakyaram Reddy, MD, Principal Investigator — Baylor Health Care System
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yadlapati R, Kahrilas PJ, Fox MR, Bredenoord AJ, Prakash Gyawali C, Roman S, Babaei A, Mittal RK, Rommel N, Savarino E, Sifrim D, Smout A, Vaezi MF, Zerbib F, Akiyama J, Bhatia S, Bor S, Carlson DA, Chen JW, Cisternas D, Cock C, Coss-Adame E, de Bortoli N, Defilippi C, Fass R, Ghoshal UC, Gonlachanvit S, Hani A, Hebbard GS, Wook Jung K, Katz P, Katzka DA, Khan A, Kohn GP, Lazarescu A, Lengliner J, Mittal SK, Omari T, Park MI, Penagini R, Pohl D, Richter JE, Serra J, Sweis R, Tack J, Tatum RP, Tutuian R, Vela MF, Wong RK, Wu JC, Xiao Y, Pandolfino JE. Esophageal motility disorders on high-resolution manometry: Chicago classification version 4.0(c). Neurogastroenterol Motil. 2021 Jan;33(1):e14058. doi: 10.1111/nmo.14058. PMID 33373111
- [Background] Richter JE, Clayton SB. Diagnosis and Management of Esophagogastric Junction Outflow Obstruction. Am J Gastroenterol. 2019 Apr;114(4):544-547. doi: 10.14309/ajg.0000000000000100. No abstract available. PMID 30848733
- [Background] Sadowski DC, Ackah F, Jiang B, Svenson LW. Achalasia: incidence, prevalence and survival. A population-based study. Neurogastroenterol Motil. 2010 Sep;22(9):e256-61. doi: 10.1111/j.1365-2982.2010.01511.x. Epub 2010 May 11. PMID 20465592
- [Background] Enestvedt BK, Williams JL, Sonnenberg A. Epidemiology and practice patterns of achalasia in a large multi-centre database. Aliment Pharmacol Ther. 2011 Jun;33(11):1209-14. doi: 10.1111/j.1365-2036.2011.04655.x. Epub 2011 Apr 11. PMID 21480936
- [Background] Okeke FC, Raja S, Lynch KL, Dhalla S, Nandwani M, Stein EM, Chander Roland B, Khashab MA, Saxena P, Kumbhari V, Ahuja NK, Clarke JO. What is the clinical significance of esophagogastric junction outflow obstruction? evaluation of 60 patients at a tertiary referral center. Neurogastroenterol Motil. 2017 Jun;29(6). doi: 10.1111/nmo.13061. Epub 2017 Apr 9. PMID 28393437
- [Background] Schupack D, Katzka DA, Geno DM, Ravi K. The clinical significance of esophagogastric junction outflow obstruction and hypercontractile esophagus in high resolution esophageal manometry. Neurogastroenterol Motil. 2017 Oct;29(10):1-9. doi: 10.1111/nmo.13105. Epub 2017 May 23. PMID 28544670
- [Background] Clayton SB, Patel R, Richter JE. Functional and Anatomic Esophagogastic Junction Outflow Obstruction: Manometry, Timed Barium Esophagram Findings, and Treatment Outcomes. Clin Gastroenterol Hepatol. 2016 Jun;14(6):907-911. doi: 10.1016/j.cgh.2015.12.041. Epub 2016 Jan 12. PMID 26792374
- [Background] Samo S, Qayed E. Esophagogastric junction outflow obstruction: Where are we now in diagnosis and management? World J Gastroenterol. 2019 Jan 28;25(4):411-417. doi: 10.3748/wjg.v25.i4.411. PMID 30700938
- [Background] Vaezi MF, Pandolfino JE, Yadlapati RH, Greer KB, Kavitt RT. ACG Clinical Guidelines: Diagnosis and Management of Achalasia. Am J Gastroenterol. 2020 Sep;115(9):1393-1411. doi: 10.14309/ajg.0000000000000731. PMID 32773454
- [Background] Nelson M, Zhang X, Genta RM, Turner K, Podgaetz E, Paris S, Cardenas J, Gu J, Leeds S, Ward M, Nguyen A, Konda V, Furuta GT, Pan Z, Souza RF, Spechler SJ. Lower esophageal sphincter muscle of patients with achalasia exhibits profound mast cell degranulation. Neurogastroenterol Motil. 2021 May;33(5):e14055. doi: 10.1111/nmo.14055. Epub 2020 Dec 6. PMID 33280206